CLINICAL TRIAL: NCT03089034
Title: Singapore Cohort of Patients with Advanced Heart Failure
Acronym: SCOPAH
Status: Active, not recruiting | Type: Observational
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: Singapore General Hospital (Other); National Heart Centre Singapore (Other)
Responsible Party: Principal Investigator, Eric A. Finkelstein, Professor, Duke-NUS Graduate Medical School
Other Study IDs: 2016/3046
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Chronic Heart Failure (CHF) is one of the leading causes of death in Singapore. Although it is well established that CHF patients in Singapore are less likely to be referred to palliative care services than cancer patients, little data is available on end-of-life (EOL) experience of advanced CHF patients in Singapore, including the inter-relationships between patient decision-making, quality of life trajectories, and health and cost consequences.

DETAILED DESCRIPTION:
To address this gap and to identify areas for better delivery of end-of-life services to patients with advanced CHF, the investigators propose to enrol a cohort of 300 patients with advanced CHF (New York Heart Association class III and IV), survey the participants every 4 months for a period of two years or till they die, whichever is earlier. The goal of this cohort study is to better understand the relationship between patient preferences, health care access, utilization, costs, and quality of life, and to identify strategies to improve the EOL experience for these patients. It is also important to recognize the significant role of the family in medical decision making in Asia. Previous studies from Singapore reveal that patients want their families to be involved in the decision making process. The role of the family in decision making is consistent with the Chinese culture of interdependency, obligations and filial piety. Decisions regarding treatment are often made by family caregivers, sometimes with little or no input from patients. Given this reality, the investigators will also enroll caregivers of the patients to evaluate their role in decision making for treatment of patients.

ELIGIBILITY:
Inclusion Criteria (patients):

* Age ≥ 21 years old
* Singaporean or Singapore Permanent Resident
* Diagnosis of advanced Congestive Heart Failure (New York Heart Association Class III and IV).
* Intact cognition (of patients ≥60 years of age) as determined by the Montreal Cognitive Assessment. If patient fails the cognitive test, he/she continues to be eligible for the study although self-reported data will no longer be collected. The primary informal caregiver of the patient will be approached for providing consent on behalf of the patient, to allow access to review of patient's medical and billing records

The inclusion criteria (primary informal caregivers)

* Age ≥ 21 years old
* Main person or one of the main providing care to the patient (e.g. accompanying patient for doctor's visits, helping the patient with day to day activities)
* Main person or one of the main ensuring provision of care (e.g. supervision of foreign domestic worker so that the patient is looked after)
* Main person or one of the main involved in making decisions regarding treatment the patient receives
* Patient they are caring for is enrolled in the study

The inclusion criteria (physicians) • Patients they are treating are enrolled in the study

Exclusion Criteria (patients):

* Patients who are not Singaporeans or Singapore Permanent Residents
* Patients who are ≤21 years of age
* Patients with psychiatric or cognitive disorders

Exclusion criteria (caregivers)

• Foreign domestic workers/ maids will be excluded from this study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced chronic heart failure(New York Heart Association class III and IV), their primary informal caregivers and their treating physicians
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-07-24 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in overall quality of life among patients through the last year of life | From recruitment to death of patient (baseline, 4 month, 8 months, 12 months, 16 months, 20 months, 24 months)
  Investigators will assess patient's quality of life through FACT-G Time frame: From recruitment to death of patient (baseline, 4 month, 8 months, 12 months, 16 months)
Change in distress among patients through the last year of life | From recruitment to death of patient (baseline, 4 month, 8 months, 12 months, 16 months, 20 months, 24 months)
  Investigators will assess patients' distress through the distress thermometer
Change in activities of daily living among patients through the last year of life | From recruitment to death of patient (baseline, 4 month, 8 months, 12 months, 16 months, 20 months, 24 months)
  Investigators will assess limitations in activities of daily living of patients through OARS Multidimensional Functional Assessment Questionnaire
Change in patient's perceived quality of care during the last year of life | From recruitment to death of patient (baseline, 4 month, 8 months, 12 months, 16 months, 20 months, 24 months)
  Investigators will describe patients' assessment of their own care using a scale used by Ayanian et al (JCO, 2010) that consists of 13 questions.
Change in patient's compliance with treatment regimens and self-care behaviours | From recruitment to death of patient (baseline, 4 month, 8 months, 12 months, 16 months, 20 months,24 months)
  Investigators will describe patients' compliance with their self-care behaviour using the Self Care of Heart Failure Index (SCHFI)
Total health care expenditure during the last year of life through analysis of medical bills | From recruitment to death of patient (baseline, 4 month, 8 months, 12 months, 16 months, 20 months, 24 months)
  Investogators will calculate total health care expenditure during the last year of patient's life as the sum total of expenditures incurred at clinics etc
Change in patients' cognitive status | From recruitment to death of patient (baseline, 4 month, 8 months, 12 months, 16 months, 20 months, 24 months)
  Investigators will assess patients' cognitive status through Montreal Cognitive Assessment

SECONDARY OUTCOMES:
Change in patient's awareness of hospice palliative care services among heart failure patients | From recruitment to death of patient (baseline, 4 month, 8 months, 12 months, 16 months, 20 months, 24 months )
  Investigators will assess change in patients' awareness of hospice palliative care services by asking them if they are aware and are using hospice palliative care services.
Change in caregiver burden through the last year of life | From recruitment to death of patient (baseline, 4 month, 8 months, 12 months, 16 months, 20 months, 24 months)
  Investigators will assess caregiver burden through modified Caregiver Reaction Assessment Scale Instrument
Change in caregiver's level of emotional distress through the last year of life | From recruitment to death of patient (baseline, 4 month, 8 months, 12 months, 16 months, 20 months, 24 months)
  Investigators will assess caregiver's anxiety and depression through the Hospital Anxiety and Depression Scale (HADS).
Caregiver's perception of patient's end-of-life care assessed after patient's death | 8 weeks bereavement
  Investigators will assess caregiver perceived quality of end-of-life care through CEQUEL.

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee JJ, Malhotra C, Sim KLD, Yeo KK, Finkelstein E, Ozdemir S. A Longitudinal Study of the Association of Awareness of Disease Incurability with Patient-Reported Outcomes in Heart Failure. Med Decis Making. 2025 Jan;45(1):97-108. doi: 10.1177/0272989X241297694. Epub 2024 Nov 15. PMID 39545423
- [Derived] Malhotra C, Foo R, Singh R, Ozdemir S, Teo I, Sim D, Jaufeerally F, Aung T, Keong YK, Nadkarni N, Finkelstein EA. Study protocol for a cohort study of patients with advanced heart failure in Singapore. BMJ Open. 2018 Sep 17;8(9):e022248. doi: 10.1136/bmjopen-2018-022248. PMID 30224389